CLINICAL TRIAL: NCT02175719
Title: Post-marketing Surveillance of Administration of Botulinum Toxin Type B(NerBloc)-Investigation of the Clinical Condition in Patients With Change From Botulinum Toxin Type A
Status: Completed | Type: Observational
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: NB02T
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Cervical Dystonia
Keywords: Torticollis; rimabotulinumtoxinB
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- E2014

SUMMARY:
Investigation of the clinical condition in patients with cervical dystonia by Toronto Western Spasmodic Torticollis Scale (TWSTRS)

ELIGIBILITY:
Inclusion criteria:

Patients with cervical dystonia who was treated by botulinum toxin type A in the past.

Patients who was enrolled in NB01S and was evaluated by TWSTRS at the first injection of NerBloc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cervical dystonia who was treated by botulinum toxin type A in the past.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-04-16 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Whole improvement level | Up to 1 year
  Toronto Western Spasmodic Torticollis Scale (TWSTRS)

CONTACTS AND LOCATIONS:
Overall Officials: Akira Endo, Study Director — Drug Fostering and Evolution Coordination Department, Eisai Co., Ltd.
Locations (2):
- Japan (2):
  - Osaka
  - Tokyo